CLINICAL TRIAL: NCT03838809
Title: Effect of a Neurological Physiotherapy Program With Electromyography-biofeedback on the Motor Activation of the Extension of the Hand and Dorsiflexion of the Foot in Cerebrovascular Damage: A Randomized Clinical Trial
Brief Title: Electromyography-biofeedback on the Motor Activation of the Extension of the Hand
Acronym: EMGBIO-ICTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Jose Hernández Morante, Principal Investigator of the Eating Disorders Research Unit, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UCAM/UITA/03
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Stroke, Complication
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION (Experimental): A group that underwent a neurological physiotherapy program with electromyography-biofeedback on the hand and the foot
  Interventions: Device: surface electromyography-biofeedback
- CONTROL (Active Comparator): A group that underwent a conventional physiotheraphy intervention
  Interventions: Device: surface electromyography-biofeedback

INTERVENTIONS:
Device: surface electromyography-biofeedback — Two electrodes were putted on the motor point of the extensor muscle of the hand and the foot. The positive electrode was placed on the distal zone of the hand or the foot, while the negative electrode was placed on the proximal zone.

SUMMARY:
Background: Biofeedback-Surface electromyography (BIO-SEMG) is a relatively recent physiotherapy technique. Although its use is widespread in sports science and sports performance, its use for the rehabilitation of patients with neurological pathologies is less studied.

Objective: The purpose of this research was to determine the changes that occur in the application of BIO-SEMG in the muscles responsible for the extension and the dorsiflexion of the hand and the foot in subjects with cerebrovascular damage.

Design: A randomized, double-blind, two-arm parallel group study was performed.

Patients: A sample of 28 subjects with limited extension of the hand and dorsiflexion of the foot as a consequence of a stroke was randomized divided in intervention or control groups.

Methods: The subjects of the intervention group underwent 12 sessions of BIO-SEMG, of 15-minute duration each of them, in the upper and lower members. On the other hand, the control group underwent another 12 sessions of 15-minute duration, in which manual physiotherapy techniques were performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a stroke
* Limitation of the hand and foot extension

Exclusion Criteria:

* Patients with some contraindication against the surface electromyography biofeedback technique, for instance, people with pacemaker, with cardiovascular antecedents, etc.
* Patients receiving other physiotherapy treatment 2 months before the beginning of the study
* Patients that decline to sign the informed consent.

Ages: 74 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Extension Degree | 3 months
  Change in the extension ability of the upper an lower members depending on the activity of the extensor muscles

SECONDARY OUTCOMES:
Fugl Meyer Test | 6 months
  Severity degree of the stroke-derived consequences

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Hernández Morante, PhD, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamez AB, Hernandez Morante JJ, Martinez Gil JL, Esparza F, Martinez CM. The effect of surface electromyography biofeedback on the activity of extensor and dorsiflexor muscles in elderly adults: a randomized trial. Sci Rep. 2019 Sep 11;9(1):13153. doi: 10.1038/s41598-019-49720-x. PMID 31511629